CLINICAL TRIAL: NCT04036175
Title: Comparison of Patient Work of Breathing and Tidal Volumes With High-flow Nasal Cannula Oxygen Therapy and Non-invasive Ventilation After Extubation in the ICU: a Prospective, Randomized, Controlled Study
Brief Title: Comparison of Patient Work of Breathing and Tidal Volumes With High Flow Nasal Cannula Oxygen Therapy and NIV (Non-Invasive Ventilation) After Extubation in the ICU.
Acronym: OVNI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A02838-45
Record Dates: First submitted 2019-06-17; First posted 2019-07-29 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: ICU; Extubation; Non-invasive Ventilation; High-Flow Nasal Oxygen Therapy; Respiratory Effort; Work of Breathing; Tidal Volume
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Standard oxygen - High-Flow Nasal Oxygen - Non-invasive ventilation - Standard Oxygen (20 minutes for each condition)
  Interventions: Device: High-Flow Nasal Oxygen / Non-invasive ventilation / Standard oxygen
- Group 2 (Other): Standard oxygen - Non-invasive ventilation - High-Flow Nasal Oxygen - Standard Oxygen (20 minutes for each condition)
  Interventions: Device: High-Flow Nasal Oxygen / Non-invasive ventilation / Standard oxygen

INTERVENTIONS:
Device: High-Flow Nasal Oxygen / Non-invasive ventilation / Standard oxygen — Device High Flow Nasal Oxygen: gas flow of 50L:Min and FiO2 adjusted to obtain SpO2>= 92% Device NIV: Pressure-support level to achieve an expired tidal volume between 6 and 8 ml/kg and PEEP level of 5 cmH2O and FiO2 adjusted for SpO2>= 92%

SUMMARY:
This study is aimed at evaluating patient work of breathing and tidal volumes with three methods of oxygenation: standard oxygen, high-flow oxygen therapy and non-invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 18 years
* planned extubation decided by the physician in charge of the patient after success of weaning trial
* patients at high risk of reintubation according to the following criteria: patient older than 65 years, or those having any underlying chronic cardiac or lung disease
* Hypoxemia defined by PaO2/FiO2 < 300 mmHg under mechanical ventilation before extubation

Exclusion Criteria:

* Duration of mechanical ventilation prior to extubation < 24h
* Contraindication to NIV
* Contraindication to nasogastric tube
* Do-not-reintubated order at time of extubation
* People under legal protection
* Opposition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2020-03-06 (Estimated); Study Completion 2020-03-06 (Estimated)

PRIMARY OUTCOMES:
Patient respiratory effort and tidal volume (Vt) | 1h20
  Swing of oesophageal pressure and pressure-Time product measured by a nasogastric pressure sensor tidal Volume estimated by electric impedance tomography

SECONDARY OUTCOMES:
Respiratory parameters | "Time 0","Time 20 min", "Time 40 min", "Time 60 min", "Time 120 min"
  respiratory rate (FR bt/min)
Respiratory parameters | "Time 0","Time 20 min", "Time 40 min", "Time 60 min", "Time 120 min"
  saturation (SpO2 in %)
Respiratory parameters | "Time 0","Time 20 min", "Time 40 min", "Time 60 min", "Time 120 min"
  transcutaneous CO2 pressure (PCO2 in mm Hg)
Respiratory parameters | "Time 0","Time 20 min", "Time 40 min", "Time 60 min", "Time 120 min"
  transpulmonary pressure (cm H2O)
Hemodynamic parameters | "Time 0","Time 20 min", "Time 40 min", "Time 60 min", "Time 120 min"
  Systolic arterial pressure (PAS in mmHg), Diastolic arterial pressure (PAD in mmHg)
Comfort evaluation | "Time 0","Time 20 min", "Time 40 min", "Time 60 min", "Time 120 min"
  comfort evaluation with an visual evaluation scale graduate 0 cm (No discomfort) to 10 cm (maximal discomfort)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud W. THILLE, PUPH, Principal Investigator — Medecine intensive reanimation CHU Poitiers
Locations (2):
- France (2):
  - CHU Poitiers, Poitiers
  - Intensive reanimation, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arrive F, Le Pape S, Bruhn A, Pepin Lehalleur A, Beuvon C, Tuffet S, Etien E, Rambault L, Frat JP, Coudroy R, Thille AW. Physiological comparison of noninvasive ventilation and high-flow nasal oxygen on inspiratory efforts and tidal volumes after extubation: a randomized crossover trial. Crit Care. 2025 May 8;29(1):185. doi: 10.1186/s13054-025-05366-y. PMID 40341100
- [Derived] Lewis SR, Baker PE, Parker R, Smith AF. High-flow nasal cannulae for respiratory support in adult intensive care patients. Cochrane Database Syst Rev. 2021 Mar 4;3(3):CD010172. doi: 10.1002/14651858.CD010172.pub3. PMID 33661521